CLINICAL TRIAL: NCT02050035
Title: Exercise and Vascular Function in Chronic Kidney Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, David Edwards, Associate Proffessor, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: KAAP32212114000; 1R01HL113514-01A1 (NIH); 364680-6 (Other: University of Delaware Institutional Review Board)
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Chronic Renal Insufficiency
Keywords: Exercise Therapy; Endothelium, vascular; Blood Vessels
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CKD Aerobic Exercise Training (Experimental): Chronic Kidney Disease participants randomly allocated to the CKD Exercise arm will receive 12 weeks of Aerobic Exercise Training three times per week.
  Interventions: Other: Aerobic Exercise Training
- CKD Control (No Intervention): Chronic Kidney Disease participants allocated to the the CKD Control arm will receive their standard routine care over a 12 week period.
- Healthy Control (No Intervention): Healthy participants will act as comparators, they will undergo baseline testing only and will not receive an intervention.

INTERVENTIONS:
Other: Aerobic Exercise Training — Supervised outpatient moderate to vigorous aerobic training at 60% - 85% heart rate reserve, carried out for 45 minutes, three times per week over a twelve week period.
  Arms: CKD Aerobic Exercise Training

SUMMARY:
The purpose of this study is to investigate the effects of 12 weeks of aerobic exercise training on blood vessel function in Stages 1-4 Chronic Kidney Disease.

DETAILED DESCRIPTION:
The endothelium lines the inside of the blood vessels. A healthy endothelial lining acts as a defense mechanism against vascular injury, mediating vascular tone, vascular structure, and blood-vessel wall relations. Endothelial dysfunction marks the occurrence of cardiovascular injuries and is a critical step in the development of cardiovascular disease. Individuals with Chronic Kidney Disease (CKD) have an increased risk of cardiovascular disease and this may be related to poor blood vessel function. Interventions to improve blood vessel function in CKD are needed. Exercise training has been shown to improve blood vessel function in older subjects and those with heart disease but this has not been investigated in CKD. The National Kidney Foundation recommends exercise for dialysis patients to reduce cardiovascular risk however there is very little data regarding the benefits of exercise in earlier stages of CKD. The purpose of this study is to determine the effect of 12 weeks of exercise training on blood vessel function in moderate to severe CKD.

ELIGIBILITY:
Inclusion Criteria:

* CKD Exercise and CKD Control Arms: Stage 1 - 4 Chronic Kidney Disease (eGFR 15 - 90 ml/min/1.73m2)
* Healthy Control Arm: eGFR > 90 ml/min/1.73m2)

Exclusion Criteria:

* History of cardiovascular disease
* Uncontrolled hypertension
* Lung disease
* Liver disease
* Cancer
* Immunosuppressant or antiretroviral therapy
* Current tobacco use
* Pregnancy
* Hormone replacement therapy
* Unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Endothelial Function | Change from baseline at 12 weeks
  Conduit artery endothelial function assessed by brachial artery flow mediated dilation; Microvascular endothelial function assessed by cutaneous vasodilation in response to local heating measured by microdialysis and laser Doppler flowmetry.

SECONDARY OUTCOMES:
Microvascular function | Change from baseline at 12 weeks
  Nitric oxide contribution to cutaneous microvascular vasodilation in response to local heating assessed by microdialysis and laser Doppler flowmetry
Oxidative stress contribution to vascular dysfunction | Change from baseline at 12 weeks
  Oxidative stress contribution to cutaneous vasodilation dysfunction in response to local heating assessed by microdialysis and laser Doppler flowmetry.
Endothelial cell oxidative stress | Changes from baseline at 12 weeks
  Endothelial cell nitrotyrosine, NADPH oxidase, MnSOD oxidase content obtained from antecubital vein endothelial cells and assessed by fluorescence microscopy.
Plasma Oxidized Low Density Lipoprotein | Change from baseline at 12 weeks
  Plasma oxidized low density lipoprotein measured by ELISA
F2-isoprostanes | Change from baseline at 12 weeks
  Urinary F2-isoprostanes measured by ELISA
Pulse Wave Analysis | Change from baseline at 12 weeks
  Central blood pressure and augmentation index assessed by oscillometry and radial tonometry
Arterial Stiffness | Change from baseline at 12 weeks
  Carotid to femoral pulse wave velocity and assessed by tonometry
Ambulatory Blood Pressure | Change from baseline at 12 weeks
  24 hour blood pressure recorded by oscillometric monitors
Peak Aerobic Capacity | Change from baseline at 12 weeks
  Peak oxygen uptake (VO2peak/max) during incremental cycling exercise until exhaustion
Physical Function | Change from baseline at 12 weeks
  Dexterity by the '9-Hole Peg Test'; Endurance by the '2 Minute Walk Endurance Test'; locomotion by the '4 Meter Gait Speed Test'; isometric handgrip strength test by handgrip dynamometry.
Habitual Physical Activity | Change from baseline at 12 weeks
  Daily average energy expenditure, step count and physical activity intensity level by accelerometry.
Knee Extensor Strength | Change from baseline at 12 weeks
  Maximal isometric knee extensor strength

CONTACTS AND LOCATIONS:
Overall Officials: David Edwards, PhD, Principal Investigator — University of Delaware
Locations (1):
- Department of Kinesiology and Applied Physiology, University of Delaware, Newark, Delaware, United States

REFERENCES:
- [Derived] Kirkman DL, Ramick MG, Muth BJ, Stock JM, Townsend RR, Edwards DG. A randomized trial of aerobic exercise in chronic kidney disease: Evidence for blunted cardiopulmonary adaptations. Ann Phys Rehabil Med. 2021 Nov;64(6):101469. doi: 10.1016/j.rehab.2020.101469. Epub 2021 Oct 26. PMID 33316435